CLINICAL TRIAL: NCT00185796
Title: Total Lymphoid Irradiation and Anti-Thymocyte Globulin as Conditioning for Non-Myeloablative Allogeneic Hematopoietic Cell Transplantation for the Treatment of Myelodysplastic Syndromes and Myeloproliferative Disorders (Except CML)
Brief Title: TLI & ATG for Non-Myeloablative Allogeneic Transplantation for MDS and MPD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Robert Lowsky, Professor of Medicine, Stanford University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMT168; 95130; BMT168; NCT00185796; 13680 (Other: Stanford IRB)
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Myeloproliferative Disorders; Blood Cancer; Myelodysplastic Syndromes
MeSH Terms: conditions — Myeloproliferative Disorders; Hematologic Neoplasms; Myelodysplastic Syndromes | interventions — Antilymphocyte Serum

ARMS (1):
- TLI/ATG conditioning (Experimental): Lymphoid irradiation and anti-thymocyte globulin (TLI/ATG).
  Interventions: Procedure: Total Lymphoid Irradiation (TLI); Procedure: Anti-Thymocyte Globulin as Conditioning (ATG)

INTERVENTIONS:
Procedure: Total Lymphoid Irradiation (TLI) — TLI is administered ten times in 120cGy fractions on day -11 through day -7 and day -4 through day -1
Procedure: Anti-Thymocyte Globulin as Conditioning (ATG) — Thymoglobulin will be administered five times intravenously at 1.5 mg/kg/day from day -11 through day -7 for a total dose of 7.5 mg/kg. Thymoglobulin doses will be based on the adjusted ideal body weight if the patient is greater than or equal to 15 kg over ideal body weight.

SUMMARY:
To evaluate the feasibility and safety of TLI/ATG conditioning for allogeneic HCT for elderly patients with advanced stage MDS and MPD.

DETAILED DESCRIPTION:
Total Lymphoid Irradiation and Anti-Thymocyte Globulin as Conditioning for Non-Myeloablative Allogeneic Hematopoietic Cell Transplantation for the Treatment of Myelodysplastic Syndromes and Myeloproliferative Disorders (except CML). To evaluate the feasibility and safety of TLI/ATG conditioning for allogeneic HCT for elderly patients or those with co-morbid conditions that preclude myeloablative transplantation for advanced stage MDS and MPD.

ELIGIBILITY:
Inclusion Criteria:

GENERAL INCLUSION CRITERIA

* General inclusion criteria must include at least one of the following:

  * Patients aged > 49 and < 75 years with MDS or MPD
  * Patients aged < 49 years at high risk for regimen related toxicity using standard high dose regimens. Factors considered high risk include pre-existing conditions such as a chronic disease affecting kidneys, liver, lungs, or heart.
  * Patients with secondary MDS following a prior autologous transplant.
* An HLA-identical related or an HLA-matched unrelated donor is available. ABO incompatibility is acceptable.
* A signed informed consent form.

MYELODYSPLASTIC SYNDROME CRITERIA

* Diagnosis of MDS classifiable by the FAB system as refractory anemia (RA), refractory anemia with ringed sideroblasts (RARS), chronic myelomonocytic leukemia (CMML), refractory anemia with excess blasts (RAEB), and MDS transformed to acute leukemia.
* Patients with advanced MDS must be cytoreduced to < 10% marrow blasts prior to receiving conditioning with TLI/ATG. Less than 10% marrow blasts must be documented by marrow examination within 1 month of starting conditioning. The cytoreductive regimen will be determined by referring centers.
* Patients with evolution to AML are required to be in a complete remission as defined by a blast count of less than 5% in a marrow aspirate with adequate cellularity. Presence of residual dysplastic features following cytoreductive therapy is acceptable.
* All patients with high risk disease, for example "intermediate-2" or "high risk" disease by the IPSS score. Other selected patients with a lower IPSS score may be considered but only after discussion with the BMT attending physicians, as a group, and the PI of the study.

MYELOPROLIFERATIVE DISORDERS

* Myeloproliferative disorders to be included:

  * Philadelphia chromosome-negative CML.
  * Patients with polycythemia vera with persistent thrombotic or hemorrhagic complications despite conventional therapy, or who have progressed to post-polycythemic marrow fibrosis.
  * Patients with essential thrombocythemia with persistent thrombotic or hemorrhagic complications despite conventional therapy, or who have progressed to myelofibrosis.
  * Patients with agnogenic myeloid metaplasia with high risk disease, for example "intermediate" or "high risk" according to the Lille Scoring System.
* Patients must be cytoreduced to < 10% marrow blasts. Less than 10% marrow blasts must be documented by marrow examination within 1 month of initiation of TLI/ATG. The cytoreductive regimen will be determined by referring centers.
* Patients with evolution to AML are required to be in a complete remission as defined by a blast count of less than 5% in a marrow aspirate with adequate cellularity. Presence of residual dysplastic features following cytoreductive therapy is acceptable.

INCLUSION CRITERIA - RELATED DONORS

* Related to the patient and is genotypically or phenotypically HLA-identical.
* Donor age < 75 unless cleared by P.I
* Capable of giving written, informed consent.
* Donor must consent to PBSC mobilization with G-CSF and apheresis

INCLUSION CRITERIA - UNRELATED DONORS

* Donors must be HLA-matched as defined by the following criteria:

  * Matched for HLA-DRB1 and DQB1 by high resolution typing.
  * Serologic match for all recognized HLA-A, HLA-B, and HLA-C antigens, and molecular match for at least 5 of 6 HLA-A, HLA-B, or HLA-C antigens by high resolution typing.
* Donor must consent to PBSC mobilization with G-CSF and apheresis. Bone marrow unrelated donors are not eligible for this protocol.

Exclusion Criteria:GENERAL EXCLUSION CRITERIA

* Organ dysfunction as defined by the following:

  * Renal: Patients with a normal creatinine are eligible for study without the need for a 24 hr urine collection for creatinine clearance. Patients with an elevated creatinine require a 24 hr urine collection. If the creatinine clearance is < 50 ml/min patients will be determined for inclusion on a case by case basis.
  * Cardiac: Ejection fraction < 40%, symptomatic congestive heart failure requiring therapy, poorly controlled cardiac arrythmias, or poorly controlled hypertension with inability to maintain a steady-state blood pressure of 150/90.
  * Pulmonary: Requirement for supplemental oxygen administration, or pulmonary function testing showing (1) DLCO < 50% of predicted, (2) TLC < 30%, or (3) FEV1 < 30%.
  * Hepatic: Patients with clinical or laboratory evidence of liver disease would be evaluated for the cause of liver disease, its clinical severity in terms of liver function and degree of portal hypertension. Patients will be excluded if they are found to have fulminant liver failure, cirrhosis if the liver with evidence of portal hypertension, alcoholic hepatitis, esophageal varices, a history of bleeding esophageal varices, hepatic encephalopathy, uncorrectable hepatic synthetic dysfunction evidenced by prolongation of the prothrombin time, ascites related to portal hypertension, bacterial or fungal liver abscess. Biliary obstruction, chronic viral hepatitis with total serum bilirubin > 3 mg/dl, and symptomatic biliary disease.
* Bone marrow documenting blast count >=10%.
* Presence of active of non-hematologic malignancy (except localized non-melanoma skin malignancies) or hematologic malignancy other than MDS or MPD as listed in inclusion criteria.
* Active CNS involvement of disease.
* Karnofsky performance score <= 60% or Lansky-Play Performance score <50 for pediatric patients.
* Life expectancy severely limited by diseases other than malignancy.
* Fungal infections with radiological progression despite with an amphotericin product or active triazole for > 1 month.
* Active bacterial infection.
* Patients of fertile age who refuse contraception for a twelve month period post-transplant.
* Pregnant or lactating females.
* HIV seropositivity.
* Severe psychological illness.

EXCLUSION CRITERIA - RELATED DONORS

* Identical twin
* Any contra-indication to the administration of subcutaneous G-CSF at a dose of 16mg/kg/d for five consecutive days
* Serious medical or psychological illness
* Pregnant or lactating females
* Prior malignancy within the preceding five years, with the exception of non-melanoma skin cancers.
* HIV seropositivity

Ages: 49 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2004-07; Primary Completion 2014-04 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
To improve survival outcome for selected patients with advanced stages of MDS and MPD with non-myeloablative allogeneic HCT from related and unrelated donors. | 7/15/2017
To evaluate the feasibility and safety of TLI/ATG conditioning for allogeneic HCT for elderly patients or those with co-morbid conditions that preclude myeloablative transplantation for advanced stage MDS and MPD. | 7/15/2017

SECONDARY OUTCOMES:
To evaluate myeloid and platelet engraftment. | 7/15/2017
To evaluate the incidence of acute and chronic GVHD. | 7/15/2017
To evaluate the rate of primary and secondary graft failure. | 7/15/2017
To evaluate the rate of relapse, survival and event-free survival. | 7/15/2017
To evaluate if DLI can be used safely in patients with mixed chimerism. | 7/15/2017

CONTACTS AND LOCATIONS:
Overall Officials: Robert Lowsky, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States